CLINICAL TRIAL: NCT02837952
Title: A Phase 3, Double-blind, Randomized Safety And Efficacy Study Comparing Multiple Administrations Of Ibu 250 Mg/Apap 500 Mg (Administered As Two Tablets Of Ibu/Apap 125 Mg/250 Mg) To Placebo In The Treatment Of Post Surgical Dental Pain In Adult Subjects
Brief Title: A Study of Ibuprofen (IBU) 250mg/APAP 500mg In The Treatment Of Post-Surgical Dental Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B5061004; GEMINI MDDP (Other: Alias Study Number); MDDP (Other: Alias Study Number)
Record Dates: First submitted 2016-05-03; First posted 2016-07-20 (Estimated); Results first posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-01

CONDITIONS: Pain
Keywords: Ibuprofen, acetaminophen, pain, molar extraction
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed Dose Combination(FDC) IBU/APAP 250 mg/500 mg (Active Comparator): FDC IBU/APAP 250 mg/500 mg
  Interventions: Drug: FDC IBU/APAP 250 mg/500 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FDC IBU/APAP 250 mg/500 mg — FDC IBU/APAP 250 mg/500 mg
  Arms: Fixed Dose Combination(FDC) IBU/APAP 250 mg/500 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is being conducted to determine the overall analgesic efficacy and safety of a fixed-dose ibuprofen 250 mg / acetaminophen 500 mg formulation compared to placebo in subjects who are experiencing post operative pain following surgical extraction of 3 or more third molar teeth. A review of any reported adverse events will also be completed.

ELIGIBILITY:
Inclusion Criteria

1. Males and females 18 years to 40 years of age (inclusive).
2. Outpatients who have undergone surgical extraction of 3 or more third molars, of which at least 2 must be a partial or complete bony mandibular impaction.
3. Subject must have at least moderate pain on the 4 point categorical scale, confirmed by at least 50 mm on the 100 mm VAS PSR scale within approximately 5 hours (ie, less than or equal to 5 hours, 15 minutes) after surgery is completed.
4. In general good health and have no contraindications to the study or rescue medication.

Exclusion Criteria

1. Presence or history of any significant hepatic, renal, endocrine, cardiovascular, neurological, psychiatric, gastrointestinal, pulmonary, hematologic, or metabolic disorder determined by the Investigator to place the subject at increased risk, including the presence or history within 2 years of screening of the following medical conditions/disorders:

   * Gastrointestinal ulcer or gastrointestinal bleeding;
   * Paralytic ileus or other gastrointestinal obstructive disorders;
   * Bleeding disorder.
2. Hypersensitivity to ibuprofen, naproxen, aspirin, or any other NSAID; or to APAP, tramadol, other opioids, or to their combinations.
3. Prior use of any type of analgesic or NSAID within five half lives of that drug or less before taking the first dose of investigational product, except for pre anesthetic medication and anesthesia for the procedure.

   .

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pharmaceutical Research Associates, Inc., Salt Lake City, Utah, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5061004&StudyName=A+Phase+3%2C+Double-blind%2C+Randomized+Safety+And+Efficacy+Study+Comparing+Multiple+Administrations+Of+Ibu+250+Mg%2Fapap+500+Mg+%28administered+As+Two+Tablets+Of+Ibu%2Fapap+125+Mg%2F250+Mg%29+To+Placebo+In+The+Treatment+Of+Post+Surgical+Dental+Pain+In+Adult+Subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to fixed dose combination of ibuprofen (IBU) / acetaminophen (APAP) (administered as 2 tablets) within 7 minutes of the completion of Baseline (0 hours on Day 1) pain assessments and, thereafter, every 8 hours up to 40 hours during the study duration of 48 hours. Participants were followed up to 28 days after the last dose of study drug (up to Day 30).
- Ibuprofen 250 mg / Acetaminophen 500 mg: Participants received fixed dose combination of IBU 250 mg/ APAP 500 mg (administered as 2 tablets of IBU 125 mg/APAP 250 mg) within 7 minutes of the completion of baseline (0 hours on Day 1) pain assessments and, thereafter, every 8 hours up to 40 hours during the study duration of 48 hours. Participants were followed up to 28 days after the last dose of study drug (up to Day 30).
Period: Overall Study
Arm/Group | Placebo | Ibuprofen 250 mg / Acetaminophen 500 mg
Started | 41 | 82
Completed | 36 | 76
Not Completed | 5 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Medication Error | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen 250 mg / Acetaminophen 500 mg | Total
Number analyzed (Participants) | 41 | 82 | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.8 (4.09) | 21.8 (3.73) | 21.8 (3.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 45 | 67
  Male | 19 | 37 | 56
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 35 | 77 | 112
  Unknown or Not Reported | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of Pain Intensity Difference Scores on 11-Point Numerical Scale From 0 to 24 Hours Post-dose (SPID11 [0-24])
Description: Pain intensity was assessed on an 11-point numerical pain severity rating scale. SPID11 [0-24]: Time-weighted sum of Pain Intensity Difference (PID) scores over 24 hours. SPID11 score range was -120 (worst score) to 240 (best score) for SPID 0-24. PID was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 =no pain to 10 =worst possible pain) from the baseline pain intensity scores (score range: 5 =moderate pain to 10 =worst possible pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID: -5 (worst score) to 10 (best score).
Time Frame: 0 to 24 hours post dose
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a Scale
Groups:
- Ibuprofen 250 mg / Acetaminophen 500: Participants received fixed dose combination of IBU 250 mg/ APAP 500 mg (administered as 2 tablets of IBU 125 mg/APAP 250 mg) within 7 minutes of the completion of baseline (0 hours on Day 1) pain assessments and, thereafter, every 8 hours up to 40 hours during the study duration of 48 hours. Participants were followed up to 28 days after the last dose of study drug (up to Day 30).
Arm/Group | Placebo | Ibuprofen 250 mg / Acetaminophen 500
Number analyzed (Participants) | 41 | 82
units on a Scale | -8.13 (9.426) | 64.76 (6.676)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg / Acetaminophen 500; Treatment difference and 95 percent (%) confidence interval (CI) were based on LS Mean from analysis of covariance (ANCOVA) with treatment, gender, baseline categorical pain severity rating (PSR) as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority; p < 0.001, ANCOVA; Least Square Mean Difference = 72.89, 95% CI 2-sided [50.075 to 95.707]

2. Secondary Outcome: Time-weighted Sum of Pain Intensity Difference Score on 11-Point Numerical Scale (SPID11) From 0 to 8, 6 to 8, 0 to 16, 8 to 16 and 0 to 48 Hours Post-dose
Description: Pain intensity was assessed on an 11-point numerical pain severity rating scale. SPID11 for various time intervals: Time-weighted sum of PID scores over time intervals of 0-8 hours, 6-8 hours, 0-16 hours, 8-16 hours and 0-48 hours. SPID11 score range was -40 (worst score) to 80 (best score) for (SPID11 [0-8]), -15 (worst score) to 30 (best score) for (SPID11 [6-8]), -80 (worst score) to 160 (best score) for (SPID11 [0-16]), -45 (worst score) to 90 (best score) for (SPID11 [8-16]), -240 (worst score) to 480 (best score) for (SPID11 [0-48]). PID was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 =no pain to 10 =worst possible pain) from the baseline pain intensity scores (score range: 5 =moderate pain to 10 =worst possible pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID: -5 (worst score) to 10 (best score).
Time Frame: 0 to 8 hours, 6 to 8 hours, 0 to 16 hours, 8 to 16 hours and 0 to 48 hours post dose
Population: The FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 250 mg / Acetaminophen 500
Number analyzed (Participants) | 41 | 82
units on a scale
  0 to 8 hours | -3.12 (2.708) | 23.33 (1.918)
  6 to 8 hours | -1.46 (1.123) | 6.45 (0.795)
  0 to 16 hours | -6.24 (6.028) | 45.43 (4.270)
  8 to 16 hours | -3.68 (3.794) | 23.64 (2.687)
  0 to 48 hours | -14.97 (19.668) | 123.69 (13.930)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg / Acetaminophen 500; 0 to 8 hours: Treatment difference and 95% CI were based on least square (LS) mean from analysis of covariance (ANCOVA) with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority; p < 0.001, ANCOVA; Least Square Mean Difference = 26.45, 95% CI 2-sided [19.895 to 33.005]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg / Acetaminophen 500; 6 to 8 hours: Treatment difference and 95% CI were based on LS mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 7.91, 95% CI 2-sided [5.196 to 10.632]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 250 mg / Acetaminophen 500; 0 to 16 hours: Treatment difference and 95% CI were based on LS mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 51.67, 95% CI 2-sided [37.075 to 66.258]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg / Acetaminophen 500; 8 to 16 hours: Treatment difference and 95% CI were based on LS mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 27.32, 95% CI 2-sided [18.139 to 36.508]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen 250 mg / Acetaminophen 500; 0 to 48 hours: Treatment difference and 95% CI were based on LS mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 138.65, 95% CI 2-sided [91.045 to 186.261]

3. Secondary Outcome: Duration of Relief After First Dose
Description: Duration of relief (in minutes) was defined as the time interval from the administration of first dose of study drug up to the administration of a rescue medication or discontinuation of the participant from the study due to lack of efficacy or administration of second dose of study drug, whichever occurred first. If prior to taking rescue medication or secondary dose, a participant discontinued early from the study due to other reasons, the time was censored at time when the participant last performed a study evaluation prior to the discontinuation.
Time Frame: Up to 8 hours after first dose
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen 250 mg / Acetaminophen 500
Number analyzed (Participants) | 41 | 82
minutes | 82.0 [75.0 to 99.0] | NA [NA to NA] — Due to less than 50% of participants who had the event, median and 95% CI was not estimable and hence not reported.
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg / Acetaminophen 500; Test type: Superiority; p < 0.001, Gehan-Wilcoxon test — P-value Method was based on Gehan-Wilcoxon test, stratified by sex and baseline categorical PSR

4. Secondary Outcome: Time to Onset of "Meaningful" Pain Relief After First Dose
Description: Using the double stopwatch method, participants started two stopwatches soon after dosing. Participants evaluated time to meaningful relief after first dose by stopping the second stopwatch labelled as "meaningful relief" at the moment they first began to experience meaningful relief after the administration of first dose and prior to the administration of second dose of study drug. The stopwatch was active for up to 8 hours after dosing or until stopped by the participant, or until second dose or a rescue medication whichever is administered first.
Time Frame: Up to 8 hours after first dose
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen 250 mg / Acetaminophen 500
Number analyzed (Participants) | 41 | 82
minutes | 165.9 [88.0 to 170.0] | 59.2 [47.7 to 74.5]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg / Acetaminophen 500; Test type: Superiority; p < 0.001, Gehan-Wilcoxon test — P-value Method was based on Gehan-Wilcoxon test, stratified by sex and baseline categorical PSR

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after the last dose (up to 30 days)
Arm/Group | Placebo | Ibuprofen 250 mg / Acetaminophen 500 mg
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/82
Other Adverse Events (participants affected / at risk) | 14/41 | 11/82
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Ibuprofen 250 mg / Acetaminophen 500 mg (N=82)
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 8 | 5
Sensitivity of teeth (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 4
Chest discomfort (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 4 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT02837952/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT02837952/SAP_001.pdf